CLINICAL TRIAL: NCT00966355
Title: RCT for the Effect of Early Administration of Vasoactive Substances When Combined With Endoscopic Treatment in Acute Gastro-esophageal Variceal Bleeds: Comparisons Among Terlipressin, Somatostatin, and Octreotide
Brief Title: Comparison of Terlipressin, Somatostatin, and Octreotide for Control of Variceal Bleeding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Soon Ho Um, Professor, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPSTOT
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2017-08

CONDITIONS: Variceal Bleeding, Cirrhosis
Keywords: Cirrhosis, Esophagus Disorders, Varicose Veins
MeSH Terms: conditions — Fibrosis; Esophageal Diseases; Varicose Veins | interventions — Terlipressin; Somatostatin; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Terlipressin (Active Comparator): treat with terlipressin IV for 5 days and endoscopic treatment
  Interventions: Drug: Terlipressin
- Somatostatin (Active Comparator): treat with somatostatin IV for 5 days and endoscopic treatment
  Interventions: Drug: Somatostatin
- Octreotide (Active Comparator): treat with octreotide IV for 5 days and endoscopic treatment
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Terlipressin — loading with 2 mg IV, and then 1 mg IV every 4 hours for 5 days
  Other Names: Glypressin
  Arms: Terlipressin
Drug: Somatostatin — loading with 250 microgram IV, and then 250 microgram/hour continuous IV for 5 days
  Other Names: Somatosan
  Arms: Somatostatin
Drug: Octreotide — loading with 50 microgram IV, and then 25 microgram/hour continuous IV for 5 days
  Other Names: Sandostatin
  Arms: Octreotide

SUMMARY:
This study is performed to compare the efficacy of terlipressin, somatostatin, and octreotide in patients with variceal bleeding for the control of variceal bleeding in combination with endoscopic therapy.

DETAILED DESCRIPTION:
In patients who are suspected to have variceal bleedings, pharmacologic therapy with vasoactive drugs such as terlipressin, somatostatin, and octreotide is recommended as soon as possible, even before endoscopy. However, it is still unclear whether the efficacies of these drugs are same or not. This study is performed to compare the efficacy of terlipressin, somatostatin, and octreotide in patients with variceal bleeding for the control of variceal bleeding in combination with endoscopic therapy.

ELIGIBILITY:
Inclusion Criteria:

* liver cirrhosis
* age between 16 and 75 years
* Patients who have upper GI bleeding symptoms (hematemesis or melena) within 24 hours before enrollment
* Patients whose systolic blood pressure <100 mmHg or pulse rate >100/min at the enrollment
* Patients who were not performed endoscopic or pharmacologic therapy for varices
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Positive anti-HIV Ab
* A history of severe side-effects or contraindications to study drugs
* Severe cardiovascular diseases: acute myocardial infarction, A-V block, congestive heart failure, ischemic heart disease, hypertension (systolic blood pressure >170 mmHg or diastolic pressure >100 mmHg)
* Chronic renal failure
* Hepatocellular carcinoma with protal vein thrombosis
* Coexisting malignancy except hepatocellular carcinoma

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1034 (Actual)
Dates: Start 2006-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soon Ho Um, Prof, Principal Investigator — Korea University
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with liver cirrhosis presenting with either hematemesis or melena between October 1, 2006 and May 31, 2010 at eleven medical centers distributed throughout Korea.
Pre-assignment Details: failure to fulfill inclusion criteria, no cirrhosis, prior endoscopic therapy within 2 weeks, enrolled within 6 weeks before index bleed, severe cardiovascular diseases, chronic renal failure, hepatocellular carcinoma invading portal vein, other malignancy, pregnancy, HIV-positive, hypersensitivity to the study drugs, or refusal to participate.
Groups:
- Octreotide: treat with octreotide IV for 5 days and endoscopic treatment
  Octreotide : loading with 50 microgram IV, and then 25 microgram/hour continuous IV for 5 days
- Somatostatin: treat with somatostatin IV for 5 days and endoscopic treatment
  Somatostatin : loading with 250 microgram IV, and then 250 microgram/hour continuous IV for 5 days
- Terlipressin: treat with terlipressin IV for 5 days and endoscopic treatment
  Terlipressin : loading with 2 mg IV, and then 1 mg IV every 4 hours for 5 days
Period: Overall Study
Arm/Group | Octreotide | Somatostatin | Terlipressin
Started | 344 | 345 | 345
Completed | 260 | 259 | 261
Not Completed | 84 | 86 | 84
Not completed — non-variceal bleeding on endoscopy | 68 | 70 | 71
Not completed — newly diagnosed advanced HCC | 11 | 12 | 10
Not completed — Lost to Follow-up | 5 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Octreotide | Somatostatin | Terlipressin | Total
Number analyzed (Participants) | 260 | 259 | 261 | 780
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 220 | 218 | 223 | 661
  >=65 years | 40 | 41 | 38 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (10.0) | 53.1 (9.7) | 52.9 (9.2) | 53.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 43 | 38 | 114
  Male | 227 | 216 | 223 | 666
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 260 | 259 | 261 | 780

OUTCOME MEASURES:

1. Primary Outcome: 5-day Treatment Failure (Failure to Control Bleeding, Rebleeding, or Death)
Time Frame: 5 days after enrollment
Measure: Number; unit: participants
Arm/Group | Octreotide | Somatostatin | Terlipressin
Number analyzed (Participants) | 260 | 259 | 261
participants | 218 | 216 | 225

2. Secondary Outcome: Active Bleeding During the First Endoscopic Exam, Needing Blood Transfusion for 5 Days, Experiencing Adverse Effects
Description: at least one of the three criteria
Time Frame: 5 days after enrollment
Measure: Number; unit: participants
Arm/Group | Octreotide | Somatostatin | Terlipressin
Number analyzed (Participants) | 260 | 259 | 261
participants | 113 | 115 | 114

ADVERSE EVENTS:
Arm/Group | Octreotide | Somatostatin | Terlipressin
Serious Adverse Events (participants affected / at risk) | 0/260 | 0/259 | 0/261
Other Adverse Events (participants affected / at risk) | 3/260 | 3/259 | 4/261
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octreotide (N=260) | Somatostatin (N=259) | Terlipressin (N=261)
diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 4 (4) — Diarrhea developed in 2 patients. Both patients were included in the octreotide group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No